CLINICAL TRIAL: NCT06416579
Title: Comparison of the Efficiency of Schroth Method and Schroth Method Based Virtual Reality Exercises in Individuals With Adolescent Idiopatic Scoliosis
Brief Title: Comparison of the Efficiency of Schroth Method and Virtual Reality Exercises in Individuals With AIS
Acronym: RCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Irem Kurt, PhD (c), Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IUC4
Record Dates: First submitted 2024-05-12; First posted 2024-05-16 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Scoliosis; Adolescence; Scoliosis; Scoliosis Lumbar Region; Adolescent Idiopathic Scoliosis
Keywords: Scoliosis; exercise; rehabilitation; Adolescent; exercise therapy; Physical Therapy Modalities
MeSH Terms: conditions — Scoliosis; Motor Activity | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group I-Schroth Exercise Group (Experimental): Participants will be given individually structured scoliosis-specific three-dimensional exercises according to the Schroth method, 2 days a week for 12 weeks, 1 day a week for the next 12 weeks, under the supervision of a physiotherapist, for a total of 36 sessions. Participants will be given a home exercise program to do on the days they do not come to the session, and will be asked whether they have done it or not when they come to each session. The exercise program will be divided into 4 phases: 0-4, 5-8, 9-12, 12-24. Progress in the exercises will be made positionally by increasing the number of repetitions and the number of rotational breathing during the exercise.
  Interventions: Other: Schroth Exercise Group
- Group II-Schroth Method Based Virtual Reality Group (Experimental): Participants will undergo a Schroth method-based virtual reality exercise program under the supervision of a physiotherapist, 2 days a week for 12 weeks, and 1 day a week for the next 12 weeks, for a total of 36 sessions. Participants will be given a home exercise program to do on the days they do not come to the session, and will be asked whether they have done it or not when they come to each session. Schroth method based virtual reality exercise program will be made on Nintendo Wii. Games within Nintendo Wii will be implemented in individually configured positions in accordance with the Schroth method.The virtual reality exercise program will be divided into 4 phases: 0-4, 5-8, 9-12, 12-24. Sessions will last 40 minutes in total, including 5 minutes of warm-up, 30 minutes of balance and sports games, and 5 minutes of cool-down. Progression will be made by difficulty level and positional in all games.
  Interventions: Other: Schroth Method Based Virtual Reality Group
- Group III-Control Group (Other): Participants in the control group will be placed on a waiting list for 24 weeks. Participants will be given initial, intermediate and final evaluations. Participants will not receive any exercise intervention for 24 weeks and will be able to continue their routine physical activities.
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Schroth Exercise Group — Exercises will be given in lying, sitting and standing positions. In each exercise, elongation of the spine will be ensured and the person will be positioned according to the type of scoliosis. Exercises will be given progressively in supine, prone, side sitting, sitting and standing positions. In each exercise, elongation of the spine will be ensured and the person will be positioned according to the upper and lower extremities. The exercise program will be divided into 4 phases: 0-4, 5-8, 9-12, 12-24. Progress in the exercises will be made positionally by increasing the number of repetitions and the number of rotational breathing during the exercise.
  Arms: Group I-Schroth Exercise Group
Other: Schroth Method Based Virtual Reality Group — During Schroth method-based virtual reality exercises, continuity in stabilization will be ensured by using external focus and muscular activation in positions appropriate to the Schroth method and in corrected posture. Sessions will last 40 minutes in total, including 5 minutes of warm-up, 30 minutes of balance and sports games, and 5 minutes of cool-down. Warm-up and cool-down will consist of aerobic games available in Nitendo wii. Balance games will consist of Penguin Slide, Soccer Heading, Table Tilt, Balance Bubble, Ski Slalom, Ski Jump, Tilt City and Snowboard Slalom. Among the sports games, Bowling, Boxing, Tennis and Baseball will be included in the program. Progression will be made by difficulty level and positional in all games. The exercises will be made more difficult by side sitting, side sitting on a stool, sitting position, knight position, standing, sitting on a balance ball, standing on a soft floor, on a bosu ball and moving towards the balance board.
  Arms: Group II-Schroth Method Based Virtual Reality Group
Other: Control Group — Participants in the control group will be placed on a waiting list for 24 weeks. Participants will not receive any exercise intervention for 24 weeks and will be able to continue their routine physical activities.
  Arms: Group III-Control Group

SUMMARY:
Adolescent idiopathic scoliosis (AIS) is a three-dimensional deformity of the spine of unknown etiology, in the treatment of which physiotherapy-specific scoliosis-specific exercise (PSSE), corset and surgical treatment approaches are used depending on the severity of the curvature [8, 9]. The Schroth method, one of the PSSE methods, has been shown to reduce the severity of the curvature, Cobb angles and the need for surgery, especially in curvatures between 10-30 degrees, slow down the progression of the curvature, increase back muscle strength and improve respiratory functions [10-12]. In the Schroth method, mental imagery, exteroceptive, proprioceptive stimulations and mirror control, which follow motor learning principles and include internal focus, are used to increase body awareness and facilitate the individual's self-posture corrections with postural, sensorimotor and rotational breathing exercises specific to scoliosis [5, 10]. In cases that require long-term treatment, such as scoliosis, the motivation and participation of the child and adolescent population in particular decreases and negatively affects the success of treatment [1, 2]. Additionally, it has been reported in the literature that patients have difficulty in performing Schroth exercises at home and adapting the corrected posture to daily life[5]. For this reason, in order to maintain the corrected posture and make it permanent, motor learning-based approaches must be used [6]. Virtual reality rehabilitation (VR) creates an external focus on the individual, allows for a large number of repetitions, and thus encourages motor learning. It is also known that VR increases motivation, participation and exercise performance in children and adolescents[7]. When the literature was examined, no studies were found regarding VR in individuals with AIS.

The study will show that Schroth-based VR will be effective on spinal parameters, trunk rotation and spinal mobility parameters in cases with AIS. Our aim is to examine the effects of Schroth-based VR in comparison with Schroth exercises in cases with AIS.

DETAILED DESCRIPTION:
Schroth method, applied in the conservative treatment of adolescent idiopathic scoliosis (AIS), uses internally focused feedback to increase body awareness and maintain corrected posture. However, it has been reported in the literature that patients have difficulty in performing exercises at home and adapting the corrected posture to daily life[5]. In addition, since scoliosis rehabilitation requires long-term follow-up, patients' participation in treatment, motivation and exercise performance decrease over time [1, 2]. Virtual reality rehabilitation (VR) creates an external focus on the individual, allows for a large number of repetitions, and thus encourages motor learning [3, 4, 6]. It is also known that SGR increases motivation, participation and exercise performance in children and adolescents[7]. When the literature was examined, no studies were found regarding SGR in individuals with AIS.

The primary aim of our study is to investigate the comparative effects of Schroth-based VR and Schroth exercises on spinal parameters, trunk rotation and spinal mobility in cases with AIS. This study's secondary aim is that these exercise trainings; To comparatively examine the effects on postural parameters, trunk isometric muscle strength, endurance, proprioception, deformity perception, quality of life and satisfaction.

H1 hypothesis: There is a difference between the effects of Schroth-based SGR and Schroth exercises on spinal parameters, trunk rotation and spinal mobility in cases with AIS.

H0 hypothesis: In cases with AIS, there is no difference between the effects of Schroth-based SGR and Schroth exercises on spinal parameters, trunk rotation and spinal mobility.

Cases that meet the inclusion criteria will be randomly divided into groups as Group I - Schroth Group, Group II - SGR Group -, Group III - Control Group, and a 24-week program will be applied. Evaluations will be performed at baseline, 12 and 24 weeks. We think that our study will be an effective, innovative, technology-based approach that will contribute to the development of spinal and postural parameters in cases with AIS.

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with Adolescent Idiopathic Scoliosis by an orthopedic specialist
* Being between the ages of 10 and 15
* Risser 0-3 stage
* The Cobb angle determined on the anteroposterior radiograph should be 10-30 degrees.
* Major curvature being lumbar curvature
* No pulmonary or rib cage-related disease such as rib fracture, atelectasis, or asthma
* Ability to understand and follow instructions
* Volunteering to participate in the study

Exclusion Criteria:

* Using a brace
* Having received any scoliosis treatment or spine surgery within the last year
* The patient has any contraindications to exercise
* Presence of neuromuscular, orthopedic, rheumatic diseases or vestibular problems that may affect balance, vision-related diseases or mental problems.
* Another exercise or physical activity that may affect trunk muscle strength or balance
* Presence of any problem that may affect walking other than scoliosis
* Patients who cannot understand and follow instructions

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Spinal Parameters | Baseline and 24th week
  The most commonly used method to measure the size of the scoliosis curve is the Cobb angle. As a standard, measurement is made on a posteroanterior spine radiograph taken while standing. To determine the boundaries of scoliosis, a line is drawn parallel to the upper line of the vertebra with the greatest deviation. Similarly, for the lower border, a line is drawn parallel to the lowest vertebra. Vertical lines parallel to these two lines are drawn and the angle between the two lines is recorded. In our study, the Cobb angle will be measured and recorded in the sagittal and frental planes, based on the same vertebral endplates, on the spine x-ray taken at the beginning and after 24 weeks of treatment by the orthopedic and traumatology physician during the routine follow-up of the patient.
Risser Sign Evaluation | Baseline and 24th week
  Risser sign is defined as the change of the pelvic growth plate from cartilage to bone. Gradual ossification of the growth plate on the iliac apophysis from anterolateral to posteromedial is evaluated. Evaluations will be determined by the orthopedic and traumatology physician during routine follow-ups of the patient based on x-rays.
Angle of Trunk Rotation Measurement | Baseline, 12th week and 24th week
  Trunk rotation angle will be measured with a Bunnell scoliometer. There is a metal sphere inside the scoliometer that moves between 0-30˚ in the water bed. Measurements will be made by placing the scoliometer vertically on the axial axis of the spine, perpendicular to the spinosus processes of the vertebra. The evaluation will be carried out standing, in a forward bending position with hands extended forward. To adjust the distance between the feet, the physiotherapist places one foot between the patient's two feet and the patient is positioned. By moving the scoliometer from the beginning of the thoracic region to the sacrum, the largest rotation angle in the major curvature will be recorded. In our study, trunk rotation angle will be measured and recorded at baseline, at week 12, and after 24 weeks of treatment.
Spinal Mobility Evaluation | Baseline, 12th week and 24th week
  Evaluation of spinal mobility was performed with a portable, computer-aided electromechanical device (the Spinal Mouse System, Idiag, Fehraltorf, Switzerland) called "Spinal Mouse" (SM). The SM is an external, non-invasive measurement device that can evaluate spinal angles and curvatures in the frontal and sagittal planes. It has been reported that SM can be used as a reliable, fast and easy-to-use measurement method with no side effects for clinical research and patient follow-up in AIS. Measurements were made between the spinous process of the 7th cervical vertebra and the top of the anal fold (approximately the level of the sacral 3rd vertebra). Maximum right-left lateral flexion degrees in the frontal plane and maximum flexion-extension degrees in the sagittal plane will be measured and recorded.

SECONDARY OUTCOMES:
Spinal proprioception assessment: | Baseline, 12th week and 24th week
  In our study, a dual inclinometer (Acumar) with an inter-individual reliability of 0.90 and an inter-test reliability of 0.85 will be used to evaluate the active repositioning sensation of the spine. Active repositioning sensation of participants' thoracic and lumbar spines; It will be measured for flexion, extension and right-left lateral flexion. In addition to these measurements in the thoracic region, right-left rotation movements will also be included in the evaluation. The absolute difference in degrees between two positions is noted as the reposition deviation value. This test is repeated 5 times for each movement. In the evaluation made before, at the 12th week and after the treatment, the average of 5 measurements will be taken and the results will be compared. The decrease in the reposition deviation value is evaluated as the improvement in the reposition feeling.
Trunk Isometric Muscle Strength | Baseline, 12th week and 24th week
  Evaluation of trunk flexion, extension and right-left lateral flexion isometric muscle strength will be performed with a manual muscle testing device, which is an objective, valid and reliable method. Trunk flexion evaluation will be performed in the 30-degree supine position, trunk extension in the prone position, and lateral flexion in the sitting position.
Trunk Muscle Endurance | Baseline, 12th week and 24th week
  Three core endurance tests created by McGill, consisting of the lateral bridge test, trunk extension test and trunk flexion test, will be evaluated. Before each test, the required test position will be explained to the participant and he/she will be asked to try the appropriate position.
Posterior Trunk Symmetry Index (POTSI) | Baseline, 12th week and 24th week
  POTSI is a valid and reliable objective method used in the evaluation of trunk asymmetry. The POTSI parameter is defined as the sum of six indices: three frontal plane asymmetry indices (C7, axilla folds, and waist lines) and three frontal plane height difference indices (acromions, axilla folds, and waist lines). The POTSI score is calculated by placing the indices in the formula on the patient's photograph taken from the posterior. The POTSI score, which indicates complete symmetry, is zero, and a higher score indicates increasing body asymmetry. In our study, SCODIAC (SCOliotic DIAgnostiCs) computer software program will be used to calculate POTSI.
Anterior Trunk Symmetry Index (ATSI) | Baseline, 12th week and 24th week
  ATSI is another valid and reliable objective method used to evaluate trunk asymmetry, and its use together with POTSI is recommended in studies. It is defined as the sum of six indices determined on the patient's anterior photograph: three frontal plane asymmetry indices (stern notch, axillary folds and waist lines) and three frontal plane height difference indices (acromions, axillary folds and waist lines). Calculation is made by placing the indices into the formula. In our study, SCODIAC (SCOliotic DIAgnostiCs) computer software program will be used to calculate ATSI.
Walter Reed Visual Assessment Scale (WRVAS) | Baseline, 12th week and 24th week
  It is a scale developed to evaluate the physical deformity perceived by patients with idiopathic scoliosis. A high score means high deformity. The scale can be completed by the patient, the person responsible for the patient's care, and the clinician performing the evaluation. In our study, this scale will be filled in by the patient.
Global Rating of Change (GRC): | Baseline, 12th week and 24th week
  GRC is used frequently in clinical research, especially in the field of the musculoskeletal system. This scale is designed to determine the extent of improvement or deterioration of the patient over time. It also indicates the effect of an intervention or the clinical course of a condition. In the GRC scale, the patient is asked to indicate the difference between his current health status and his health status before a specific point in time. The questions asked, the number of points on the scale, and the labels assigned to the scale points may vary [29]. A 7-point scale (-3: much worse, -2: worse, -1: slightly worse, 0: the same, 1: slightly better, 2: quite better, 3: much better) will be used in our study.
"Scoliosis Research Society Scale-22 (SRS-22)" | Baseline, 12th week and 24th week
  SRS-22 is a scoliosis-specific quality of life questionnaire with 22 questions and five subgroups. Subgroups of the survey; pain, image/appearance, function/activity, mental health and treatment satisfaction. It is defined as 0 (worst) and 5 (best) points for each question. The form will be filled out by asking patients to mark the answers that apply to them. If they do not understand the questions, the questions will be explained and the answers will be marked.

CONTACTS AND LOCATIONS:
Overall Officials: İrem KURT ULUSOY, PhD(C), Principal Investigator — Istanbul University - Cerrahpasa
Locations (1):
- İrem Kurt, Istanbul, Turkey (Türkiye)